CLINICAL TRIAL: NCT02478385
Title: Birth Environment of the Future - a Randomised Controlled Study
Brief Title: Birth Environment of the Future
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herning Hospital (Other)
Responsible Party: Principal Investigator, Iben Lorentzen, Midwife, Master in Health Hummanities (MHH), Herning Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: fremtidensfødemiljø
Record Dates: First submitted 2015-03-17; First posted 2015-06-23 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy
Keywords: Birth environment; oxytocin; epidural; analgesia; home-like
MeSH Terms: conditions — Agnosia | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Birth environment labour room (Active Comparator): Supportive care of labour room designed with special attention on sound and light effects, covering medical devices and insulation from outside noise
  Interventions: Other: Supportive care in a specially designed labour room
- Labour in a standard labour room (Placebo Comparator): The woman gives labour in a standard labour room
  Interventions: Other: Supportive care in a specially designed labour room

INTERVENTIONS:
Other: Supportive care in a specially designed labour room — Light and sound effects, homelike design in furniture and wall paper, sound insulation of walls, covering medical devices in walls, apparatus, and cupboards

SUMMARY:
The main purpose of this study is to explore the impact of the birth environment on women's birth experience and relevant birth outcomes in the experimental Labour room compared to a standard Labour room.

DETAILED DESCRIPTION:
In the last decade, there has been an increased interest in exploring the impact of the birth environment on midwifery practice and the women's birth experiences. Results from these studies show that a home-like birth environment has positive effects on both midwifery practice and the birth experience. The hormone oxytocin that causes contractions during labour may play an important role in this context. The hormone is released when being in a safe, secure and confident environment. Therefore, it is a reasonable assumption that the birth environment also has an impact on birth outcomes.

To investigate this assumption one traditional labour room was transformed to an experimental labour room. The design of the room is inspired by knowledge from evidence-based healthcare design, which describes bringing nature into the room. Furthermore, it is possible for the parents to design their own birth setting by choosing atmosphere through sound, light and nature scenes.

ELIGIBILITY:
Inclusion Criteria:

* primiparas with a singleton pregnancy
* Gestational age 37-42
* speaks and understands Danish

Exclusion Criteria:

* Inducted delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 680 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
No. of women receiving oxytocin stimulation during Labour | From allocation at delivery ward (date, hour and minute) to delivery (date, hour, minute). Duration is recorded time in hours and minutes
  No of women augmented with oxytocin drip. The intervention is registered in the electronic patient journal. The duration in time (date,hours,minutes) of oxytocin treatment is registered in the electronic journal log

SECONDARY OUTCOMES:
Duration of labour | From allocation at delivery ward (date, hour and minute) to delivery (date, hour, minute). Duration is recorded time in hours and minutes
  Minutes of stay in labour room until delivery is registered in separate data sheet with time of arrival and time of delivery
Pain relieving interventions | From allocation at delivery ward (date, hour and minute) to delivery (date, hour, minute). Duration is recorded time in hours and minutes
  Interventions with epidural and pudendal analgesia are registered in the electronic patient journal

OTHER OUTCOMES:
Evaluation of woman-centred care during labour and childbirth | Six weeks after delivery a questionaire is e-mailed to the women
  Woman-centred care during labour and childbirth questionnaire
Paternal evaluation of the labour room environment | Two weeks after delivery a questionnaire is e-mailed to the father
  Questionaire in process of making

CONTACTS AND LOCATIONS:
Overall Officials: Iben Lorentzen, Midwife, Principal Investigator — Department of Gynecology and Obstetrics at Herning, Denmark; Finn F Lauszus, MD, Study Chair — Department of Gynecology and Obstetrics at Herning, Denmark
Locations (1):
- Department of gynaecology and obstetrics, Herning Hospital, Herning, Denmark

REFERENCES:
- [Background] Overgaard C, Fenger-Gron M, Sandall J. The impact of birthplace on women's birth experiences and perceptions of care. Soc Sci Med. 2012 Apr;74(7):973-81. doi: 10.1016/j.socscimed.2011.12.023. Epub 2012 Jan 28. PMID 22326105
- [Background] Foureur M, Davis D, Fenwick J, Leap N, Iedema R, Forbes I, Homer CS. The relationship between birth unit design and safe, satisfying birth: developing a hypothetical model. Midwifery. 2010 Oct;26(5):520-5. doi: 10.1016/j.midw.2010.05.015. Epub 2010 Aug 7. PMID 20692742
- [Background] Hodnett ED, Downe S, Edwards N, Walsh D. Home-like versus conventional institutional settings for birth. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD000012. doi: 10.1002/14651858.CD000012.pub2. PMID 15674867
- [Derived] Lorentzen I, Andersen CS, Jensen HS, Fogsgaard A, Foureur M, Lauszus FF, Nohr EA. Study protocol for a randomised trial evaluating the effect of a "birth environment room" versus a standard labour room on birth outcomes and the birth experience. Contemp Clin Trials Commun. 2019 Feb 15;14:100336. doi: 10.1016/j.conctc.2019.100336. eCollection 2019 Jun. PMID 30886935